CLINICAL TRIAL: NCT03779308
Title: Effect of Whole Body Vibration Therapy on Tone Abnormalities and Functional Abilities in Individuals With Dystonia Cerebral Palsy- a Pilot Study
Brief Title: Whole Body Vibration for Dystonia Cerebral Palsy
Acronym: WBVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-YBPA
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy; Dystonia
Keywords: whole body vibration therapy; cerebral palsy; dystonia; functional abilities; tone abnormalities
MeSH Terms: conditions — Cerebral Palsy; Dystonia

STUDY DESIGN:
Intervention Model Description: Before and after cohort study with sample size less than 20
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The participants will receive whole body vibration therapy while standing with hand support on a vibration platform.
  Interventions: Device: whole body vibration therapy

INTERVENTIONS:
Device: whole body vibration therapy — The study participants will receive the WBVT when standing still on a vibration platform independently or with own hand support on the platform rail. The vibration protocol is modified from the study by Gusso et al (2016). The WBVT training is of 20 Hertz, a peak-to-peak amplitude of 2 mm and peak acceleration of 15.79m/s or 1.61g. The sessions will be 18 minutes in length, 4 days per week for 4 weeks. The vibration frequency, duration and amplitude will be progressively increased over 2 weeks to the desired parameters.

SUMMARY:
Health bones allow us to move and walk freely without pain. Physical activities have been shown to relate to healthy bone growth. Children with physical disabilities are not able to do the same amount of exercises as their healthy peers. They are vulnerable to poor bone health, bone pain, and at high risk of osteopenia or even broken bones. This problem will extend to their adulthood.

Recently, whole body vibration therapy (WBVT) has been proven to improve bone health and muscle function in healthy adults and post-menopausal women. Promising results have been shown on gross motor skills, balance and muscle strength for children and young adults with mild cerebral palsy (CP). Most of the vibration protocols require the participants perform some simple exercises on the vibration platform.

Very limited studies have been done on children and young adults with moderate CP and almost none solely on individuals with dystonia CP. We do not know if the effect of the WBVT on individuals with dystonia CP would be the same as those with spastic CP and on those with moderate CP as those with mild CP. We also do not know if static standing on the vibration platform would have similar effects on tone abnormalities, balance and gross motor skills as doing simple exercises on the vibration platform because children and young adults with dystonia CP may not be able to freely do simple exercises on the vibration platform without extra support.

The present pilot study is to systematically investigate the effects of WBVT on tone abnormalities, balance and functional abilities in children and young adults with dystonia CP.

DETAILED DESCRIPTION:
Muscle contractions during normal movements and regular exercises are believed to build strong bones or good bone health. Children with cerebral palsy (CP), especially those with moderate severity, are unable to perform the required amount of exercise to improve their bone health as their typically developing counterparts. As a result, non-traumatic fractures and bone pain are common in children with moderate to severe CP. This problem extends to their adulthood, causing osteopenia or osteoporosis.

Whole body vibration therapy (WBVT) has been recently proven to improve bone health and muscle function in healthy adults, post-menopausal women and individuals with mild to moderate severity of CP. It has been postulated that the vibration can stimulate the muscle spindles and elicit consistent muscle contractions. This would be a great advantage to the individuals with moderate severity of CP, who have limited control in their body movements and prevent them to perform regular exercises as the normal individuals. Among the research of the WBVT for children with CP, promising results have been shown on gross motor function, balance and muscle strength for children with mild disability. Most of the studies, which yielded positive results, required the study participants to perform simple exercises on the vibration platform as the intervention. Very limited studies have been conducted on children and young adults with moderate severity of CP and almost no study solely on individuals with dystonia CP. Other than this lack of knowledge on this sub-group of CP, there are other knowledge gaps of this potential intervention to improve bone health for individuals with CP. Firstly, we do not know if the effect of WBVT on this population group would be similar or more effective than those with mild CP in terms of their tone abnormalities, gross motor function and balance, because the moderate group is greatly compromised in their mobility and extent of regular exercises when compared with those with mild CP. Secondly, preliminary results of the WBVT are promising in children and young adults with moderate severity of spastic CP. However, we do not know if these promising effects will be similar to those with dystonia or spastic dystonia CP because the vast differences in their tone and movement patterns. This pilot study aims to fill in these knowledge gaps and examine the effect of WBVT on children and young adults with moderate severity of dystonia CP in terms of muscle tone, balance and functional motor abilities.

Methods A convenience sample of 5 children and adolescents aged between 6 to 17 years and 5 young adults aged between 18 to 45 years with dystonia or spastic dystonia CP will be recruited. As this is a pilot study, we recruit mild to moderate severity of CP, i.e. Gross Motor Function Classification System (GMFCS) levels I to IV. In general, individuals of levels I and II ambulate unaided and are able to perform more advanced motor skills such as running and jumping with limitations. Individuals of level III mobilise with hand-held mobility devices such as crutches or walking frames. Individuals of levels IV have very limited functional mobility and are mostly limited to an indoor environment. Individuals with level V are non-ambulatory or totally rely on wheeled mobility aids in all environment settings.

The presence of dystonia in the recruited participants will be firstly confirmed using the Hypertonia Assessment Tool (HAT). It is a reliable and valid clinical tool to confirm the presence of dystonia in individuals with CP. Only those confirmed with dystonia or spastic dystonia CP will be included in this study. Assessments will be performed at baseline and at completion of the intervention to examine the functional abilities of the study participants.

The study participants will receive the WBVT when standing still on a vibration platform independently or with own hand support on the platform rail. The vibration protocol is modified from the study by Gusso et al (2016) and has also been tested in a pilot study by PI on a group of children, adolescents and young adults with spastic CP. The WBVT training is of 20 Hertz, a peak-to-peak amplitude of 2 mm and peak acceleration of 15.79m/s or 1.61g. The sessions will be 18 minutes in length, 4 days per week for 4 weeks. The vibration frequency, duration and amplitude will be progressively increased over 2 weeks to the desired parameters.

The study results will be presented as means and standard deviations. Due to the small sample size, non-parametric Wilcoxon Signed Ranks test will be used to compare the results before and after the WBVT. The statistical significance level is set at p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 17 years or 18 to 40 years
* With a diagnosis of CP or similar phenotype of childhood onset disability
* Presence of dystonia in their tone abnormalities
* Able to stand for 3 minutes independently or with own hand support on rails
* Able to follow simple instructions
* Able to undertake clinical examination; and
* With informed consent by the participant's parent/ guardian or participants if able

Exclusion Criteria:

* There is a history of fracture within 8 weeks of enrolment of the present study and acute thrombosis, muscle or tendon inflammation, renal stones, discopathy or arthritis as reported by their parent/ guardian or themselves if able.
* Females during pregnancy
* Metal implants in their spine and/or lower limbs

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure 66 Item Set (GMFM-66 IS) | 4 weeks
  assess gross motor function of participants

SECONDARY OUTCOMES:
Two-minute walk test (2MWT) | 4 weeks
  assess submaximal exercise capacity of participants by measuring the self-chosen pace walking distance covered in 2 minutes
Barry-Albright Dystonia Scale (BADS) | 4 weeks
  assess the severity of dystonia in a scale of 0 (no dystonia) to 4 (severe dystonia more than 50% of the time and/or prevent normal daily function). The grading will be done according to the published guidelines.Total score will be used as reported results for all the participants.
Timed up and go test | 4 weeks
  assess balance and functional mobility. The duration of the participant to complete the test task in terms of seconds will be used.
Edinburgh Visual Gait Score | 4 weeks
  assess any changes in the walking pattern in terms of 17 gait parameters in a scale of 0 (normal) to 2 (marked deviation from normal) according to the published guidelines. Total score will be used as reported results for all the participants.
Chinese version of the Pediatric Evaluation of Disability Inventory (PEDI) | 4 weeks
  assess functional capacities in the domains of daily activities, mobility and social/cognitive function. The raw scores of each domain will be used for analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Tamis W Pin, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apkon SD. Osteoporosis in children who have disabilities. Phys Med Rehabil Clin N Am. 2002 Nov;13(4):839-55. doi: 10.1016/s1047-9651(02)00026-8. PMID 12465563
- [Background] Sheridan KJ. Osteoporosis in adults with cerebral palsy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:38-51. doi: 10.1111/j.1469-8749.2009.03432.x. PMID 19740209
- [Background] van den Berg-Emons HJ, Saris WH, de Barbanson DC, Westerterp KR, Huson A, van Baak MA. Daily physical activity of schoolchildren with spastic diplegia and of healthy control subjects. J Pediatr. 1995 Oct;127(4):578-84. doi: 10.1016/s0022-3476(95)70115-x. PMID 7562279
- [Background] Mergler S, Evenhuis HM, Boot AM, De Man SA, Bindels-De Heus KG, Huijbers WA, Penning C. Epidemiology of low bone mineral density and fractures in children with severe cerebral palsy: a systematic review. Dev Med Child Neurol. 2009 Oct;51(10):773-8. doi: 10.1111/j.1469-8749.2009.03384.x. Epub 2009 Jul 8. PMID 19614941
- [Background] Henderson RC, Gilbert SR, Clement ME, Abbas A, Worley G, Stevenson RD. Altered skeletal maturation in moderate to severe cerebral palsy. Dev Med Child Neurol. 2005 Apr;47(4):229-36. doi: 10.1017/s0012162205000459. PMID 15832545
- [Background] Henderson RC, Kairalla JA, Barrington JW, Abbas A, Stevenson RD. Longitudinal changes in bone density in children and adolescents with moderate to severe cerebral palsy. J Pediatr. 2005 Jun;146(6):769-75. doi: 10.1016/j.jpeds.2005.02.024. PMID 15973316
- [Background] Rauch F. Vibration therapy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:166-8. doi: 10.1111/j.1469-8749.2009.03418.x. PMID 19740225
- [Background] Matute-Llorente A, Gonzalez-Aguero A, Gomez-Cabello A, Vicente-Rodriguez G, Casajus Mallen JA. Effect of whole-body vibration therapy on health-related physical fitness in children and adolescents with disabilities: a systematic review. J Adolesc Health. 2014 Apr;54(4):385-96. doi: 10.1016/j.jadohealth.2013.11.001. Epub 2014 Jan 1. PMID 24388109
- [Background] Saquetto M, Carvalho V, Silva C, Conceicao C, Gomes-Neto M. The effects of whole body vibration on mobility and balance in children with cerebral palsy: a systematic review with meta-analysis. J Musculoskelet Neuronal Interact. 2015 Jun;15(2):137-44. PMID 26032205
- [Background] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Background] Jethwa A, Mink J, Macarthur C, Knights S, Fehlings T, Fehlings D. Development of the Hypertonia Assessment Tool (HAT): a discriminative tool for hypertonia in children. Dev Med Child Neurol. 2010 May;52(5):e83-7. doi: 10.1111/j.1469-8749.2009.03483.x. PMID 20540176
- [Background] Pin TW, Choi HL. Reliability, validity, and norms of the 2-min walk test in children with and without neuromuscular disorders aged 6-12. Disabil Rehabil. 2018 Jun;40(11):1266-1272. doi: 10.1080/09638288.2017.1294208. Epub 2017 Mar 3. PMID 28637155
- [Background] Barry MJ, VanSwearingen JM, Albright AL. Reliability and responsiveness of the Barry-Albright Dystonia Scale. Dev Med Child Neurol. 1999 Jun;41(6):404-11. doi: 10.1017/s0012162299000870. PMID 10400175
- [Background] Fosang AL, Galea MP, McCoy AT, Reddihough DS, Story I. Measures of muscle and joint performance in the lower limb of children with cerebral palsy. Dev Med Child Neurol. 2003 Oct;45(10):664-70. doi: 10.1017/s0012162203001245. PMID 14515937
- [Background] Chen KL, Hsieh CL, Sheu CF, Hu FC, Tseng MH. Reliability and validity of a Chinese version of the Pediatric Evaluation of Disability Inventory in children with cerebral palsy. J Rehabil Med. 2009 Mar;41(4):273-8. doi: 10.2340/16501977-0319. PMID 19247548
- [Background] Williams EN, Carroll SG, Reddihough DS, Phillips BA, Galea MP. Investigation of the timed 'up & go' test in children. Dev Med Child Neurol. 2005 Aug;47(8):518-24. doi: 10.1017/s0012162205001027. PMID 16108451
- [Background] Del Pilar Duque Orozco M, Abousamra O, Church C, Lennon N, Henley J, Rogers KJ, Sees JP, Connor J, Miller F. Reliability and validity of Edinburgh visual gait score as an evaluation tool for children with cerebral palsy. Gait Posture. 2016 Sep;49:14-18. doi: 10.1016/j.gaitpost.2016.06.017. Epub 2016 Jun 15. PMID 27344448
- [Background] Gusso S, Munns CF, Colle P, Derraik JG, Biggs JB, Cutfield WS, Hofman PL. Effects of whole-body vibration training on physical function, bone and muscle mass in adolescents and young adults with cerebral palsy. Sci Rep. 2016 Mar 3;6:22518. doi: 10.1038/srep22518. PMID 26936535